CLINICAL TRIAL: NCT04167267
Title: A Randomized, Open-label, Single Dose Study to Evaluate the Safety and Pharmacokinetics of DWP14012 Tablet A and DWP14012 Tablet B in Healthy Volunteers
Brief Title: Pharmacokinetics and Safety of DWP14012 Tablet A and Tablet B in Healthy Volunteers (II)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW_DWP14012102
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Tablet B - Tablet A) (Experimental): Period 1 : DWP14012 tablet B Period 2: DWP14012 tablet A
  Interventions: Drug: DWP14012 tablet A; Drug: DWP14012 tablet B
- Sequence 2 (Tablet A - Tablet B) (Experimental): Period 1 : DWP14012 tablet A Period 2: DWP14012 tablet B
  Interventions: Drug: DWP14012 tablet A; Drug: DWP14012 tablet B

INTERVENTIONS:
Drug: DWP14012 tablet A — Period 1: DWP14012 tablet B Period 2: DWP14012 tablet A
Drug: DWP14012 tablet B — Period 1: DWP14012 tablet A Period 2: DWP14012 tablet B

SUMMARY:
This is a randomized, open-label, single dose study to evaluate the safety and pharmacokinetics of DWP14012 tablet A and DWP14012 tablet B in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged between 19 and 45 at screening
* Those whose weight is 55 kg and more and BMI is between 17.5 and 30.5 kg/m2
* Subjects who are adequate to be subjects in this study upon judgment of the investigator after physical examination, clinical laboratory test, examination by interview, etc

Exclusion Criteria:

* Subjects who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* Subjects who have gastrointestinal diseases or past history of gastrointestinal diseases (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux, Crohn's disease etc.) that may affect safety and pharmacokinetic/pharmacodynamic evaluation of study drug, and those who have past history of gastrointestinal surgery (however, except simple ppendectomy and herniotomy)
* Subjects who showed positive result for Helicobacter pylori test
* Subjects with serum AST (SGOT) or ALT (SGPT) level >1.5 times the upper limit of the normal range at the time of the screening examination
* Subjects with a history of drug abuse or a positive urine screening for drug abuse
* Subjects who have participated and taken investigational drug in any other clinical trial (including bioequivalence study) within six months prior to study drug administration
* Subjects who have donated a unit of whole blood within two months or blood components within one month prior to study drug administration

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
AUCt: Area under the drug concentration-time curve from time 0 to tau (dosing interval) | 0 hour (pre-dose), 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour
  each period
Cmax: Peak concentration of DWP14012 | 0 hour (pre-dose), 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour
  each period

SECONDARY OUTCOMES:
AUCinf: Area under the drug concentration-time curve from time 0 to infinity | 0 hour (pre-dose), 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour
  each period
Tmax: Time of maximum concentration | 0 hour (pre-dose), 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour
  each period
t1/2: Terminal elimination half-life | 0 hour (pre-dose), 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour
  each period
CL/F: Apperent Clearance | 0 hour (pre-dose), 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour
  each period
Vd/F: Apparent volume of distribution | 0 hour (pre-dose), 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 6 hour, 8 hour, 12 hour, 24 hour, 48 hour
  each period

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No